CLINICAL TRIAL: NCT04693013
Title: Use Of Virtual Reality To Reduce Anxiety And Pain During Repair Of Perineal Laceration
Brief Title: Use Of Virtual Reality To Reduce Anxiety And Pain During Repair Of Perineal Laceration And Episiotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, David Peleg, staff physician, Ziv Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0103-20-ZIV
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Perineum; Injury; Episiotomy Wound; Anxiety
MeSH Terms: conditions — Wounds and Injuries; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): use of virtual reality (VR)
  Interventions: Device: Virtual Reality for Anxiety Reduction
- Control (No Intervention): no use of VR

INTERVENTIONS:
Device: Virtual Reality for Anxiety Reduction — Virtual Reality for Anxiety Reduction during suturing of perineum
  Arms: Interventional

SUMMARY:
Virtual Reality will be used to decrease anxiety and pain during suturing of episiotomy and perineal lacerations

DETAILED DESCRIPTION:
Perineal lacerations and episiotomies are common after vaginal birth. Surgical repair of these conditions can cause discomfort and anxiety for the post-partum woman.

The purpose of this research is to determine if the use of virtual reality (VR) during repair of a perineal laceration or episiotomy can decrease the anxiety level of the woman. Other parameters that will be measured will be vital signs, time of procedure, and pain level.

84 eligible healthy women after spontaneous or instrumental vaginal birth will be enrolled. Allocation will be randomized by previous sealed envelopes. 42 in the VR group and 42 in the control group. The 42 women in the VR group will have the device placed band in use before the onset of the procedure. Anxiety level will be measured post-procedure by (STAI) State Inventory Anxiety Trait. Pain will be measure by VAS.

Assuming a significant anxiety level of 60% in women undergoing repair of a perineal laceration of episiotomy, in order to demonstrate a reduction to 30% in women using VR with a power of 80% and alpha of 0.05, 42 women will be needed in each group.

ELIGIBILITY:
Inclusion Criteria:

* Post-partum vaginal delivery, spontaneous or instrumental
* Episiotomy or 1st or 2nd degree perineal tear
* informed consent

Exclusion Criteria:

* Cesarean delivery
* 3rd or 4th degree perineal tear
* no informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety Level | Immediately after procedure
  questionairre

SECONDARY OUTCOMES:
Pain Level | Immediately after procedure
  questionairre

CONTACTS AND LOCATIONS:
Locations (1):
- David Peleg, Safed, Israel